CLINICAL TRIAL: NCT05404854
Title: Changes in Physical Activity, Sedentary Behavior and Associated Motivations Following a Rehabilitation Program for Chronic Low Back Pain Patients
Brief Title: Evolution of Physical Activity, Sedentary Behavior and Associated Motivations After Rehabilitation for Chronic Low Back Pain Patients
Acronym: LOMB'ACTIV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/MH-01; 2022-A00549-34 (Other: ANSM)
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain
Keywords: rehabilitation; sedentary; motivation; physical activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic low back pain patients: Physical Activity by wearing an accelerometer for 7 days before and after the rehabilitation program sedentarity by wearing an accelerometer for 7 days before and after the rehabilitation program Measurement of explicit motivation Measurement of implicit attitudes
  Interventions: Other: Physical Activity; Other: sedentarity; Other: Measurement of explicit motivation; Other: Measurement of implicit attitudes

INTERVENTIONS:
Other: Physical Activity — wearing an accelerometer for 7 days before and after the rehabilitation program
Other: sedentarity — wearing an accelerometer for 7 days before and after the rehabilitation program
Other: Measurement of explicit motivation — Explicit motivation will be assessed using self-report questionnaires. Explicit attitudes using a 7-point bipolar response scale, participants will be asked to indicate for each of the 4 pairs of positive and negative adjectives used how much they associate them with regular PA and sedentary behaviors, respectively. Perceived behavioral control using a 7-point bipolar response scale, patients will be asked to indicate how well they felt they were able to engage in regular PA, and limit their sedentary behaviors, respectively, based on two items. Intentions using a 7-point bipolar response scale, patients will be asked to indicate how much they intend to adopt regular physical activity, and limit their sedentary behaviors, respectively, according to two items. Fears and beliefs related to physical activity and work will be measured by the FABQ in its French version
Other: Measurement of implicit attitudes — Implicit attitudes will be assessed by administering an Implicit Association Test on physical and sedentary activities. Sitting in front of a computer, participants will see a series of words appear in the middle of the screen referring to 4 conceptual categories - located at the top of the screen. Two represent the targeted behaviours (here, physical activity versus sedentary lifestyle) while the remaining two represent attributes (here, positive versus negative adjectives). The adjectives used will be the same as those used to measure explicit attitudes. The instructions given to the participant are to classify the words as quickly as possible, according to the semantic category to which they belong

SUMMARY:
IIn 2016, chronic low back pain (CLBP) was the leading cause of years lived with disability worldwide. This condition impacts social interactions, work life, and can lead to an altered quality of life for patients.

For these patients, physical activity (PA) can reduce pain, improve function and the rate of return to work. According to the French National Authority for Health, it is the main treatment in the management of these patients. Nevertheless, the literature reports PA levels that are relatively comparable to those of the general population. Considering that a large proportion of adults struggle to meet these thresholds, we can infer that the same is true for CLBP patients. In addition to PA, the World Health Organization recommends that all adults should limit the amount of time spent in sedentary behaviors. Thus, CLBP patients should adopt an active lifestyle, characterized by regular PA and limited sedentary behaviors (SB).

In view of these elements, it is essential to implement dedicated interventions. The literature reports mixed results with work focused on PA promotion. No study has focused on i) the reduction of CS, ii) the rehabilitation programs (RP) proposed in France.

On the other hand, there is a need to better understand what determines engagement in such behaviors. Among these determinants are several psychological variables related to behavioral intentions. A recent line of research indicates that beyond these motivational dimensions, which are explicit in nature, certain implicit processes are significantly associated with the adoption or non-adoption of certain health-related behaviors. This result has been observed in the context of chronic disease (respiratory patients, metabolic patients) but remains unexplored in patients with chronic low back pain.

The aim of this study is to simultaneously question these different aspects: the effects of a RP on changes in PA and CS, in relation to motivational changes in a population of CLBP patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a rehabilitation program,
* Presenting chronic low back pain (i.e., > 3 months),
* Age > 18 years,
* Literacy.

Exclusion Criteria:

* Inability or refusal to answer a questionnaire,
* Protected adults,
* Participation in another study
* Withdrawal of consent,
* If deemed necessary by the principal investigator for the welfare and/or safety of the participant,
* In the event of an occurrence of a non-inclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited before their stay in the Physical Medicine and Rehabilitation departments of the University Hospital Centres of Clermont-Ferrand, Montpellier and Nîmes, on a voluntary basis, after medical advice and after verification of all the criteria mentioned below.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Physical Activity (PA) | between baseline to 3 months
  Change in the proportion of participants meeting the recommended PA level from pre-program (T0) to 3 months after returning home (T3) (Canning & Hicks, 2020; Ormel et al., 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (3):
- France (3):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

REFERENCES:
- [Result] Haas M, Boiche J, Tavares-Figuereido I, Courbis AL, Dupeyron A. Changes in physical activity, sedentary behaviors, and associated motivation after multidisciplinary rehabilitation program for chronic low back pain patients. Int J Rehabil Res. 2025 Jun 1;48(2):106-112. doi: 10.1097/MRR.0000000000000667. Epub 2025 Apr 9. PMID 40327431